CLINICAL TRIAL: NCT03325634
Title: A Phase I Study of Stereotactic Body Radiation Therapy for Patients With Limited Locoregional Recurrences of Ovarian and Uterine Serous Carcinoma
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Recurrent Primary Ovarian or Uterine Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1333.cc; NCI-2017-01888 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Endometrial Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo Stereotactic Body Radiation Therapy (SBRT) every other day for 3 fractions.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial studies the side effects and best dose of stereotactic body radiation therapy in treating patients with ovarian or uterine cancer that has come back. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue.

DETAILED DESCRIPTION:
This is a phase I study with a primary objective to determine maximum tolerated dose (MTD) of 3 fraction stereotactic body radiation therapy (SBRT) for abdominopelvic recurrences of ovarian cancer (OC) and uterine papillary serous carcinoma (UPSC). This is a dose escalation study that employs a 3+3 design to determine the MTD. Patients are then monitored closely to determine side effects and adverse events, as well as success rates and tumor response to the radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients > 18 years of age.
* ECOG 0 or 1.
* Diagnosis of primary ovarian cancer of any histology (patients with diagnoses of fallopian tube and primary peritoneal cancer are also eligible), or primary uterine cancer of papillary serous histology.
* Pathologic confirmation of eligible histology.
* Three or fewer total sites of active disease (at least one site of active disease to be treated on study must be confined to the abdomen or pelvis excluding liver and must be < 5 cm in greatest dimension as determined by pre-screening cross-sectional imaging).
* Additional site(s) of active disease (such as parenchymal liver and lung metastases, or supraclavicular nodal metastases), should be considered for treatment (off study) with radiation, surgery, or another form of local therapy, at the discretion of the study PI.
* Systemic therapy is allowed but SBRT cannot begin until > or = 7 days after the last cycle of systemic therapy, and systemic therapy cannot be initiated or re-initiated until > or = 7 days after SBRT. There will be no limit on prior lines of systemic therapy.
* Patients with contraindications to intravenous (IV) contrast administration are still eligible for this study if the tumor can be delineated clearly without IV contrast (at the discretion of the treating radiation oncologist) but will not participate in the functional imaging studies.

Exclusion Criteria:

* Pregnant women. If patients are not status post bilateral salpingo-oopherectomy then pregnancy testing is required.
* Patients with active collagen vascular disease (CVD), specifically systemic lupus erythematosus or scleroderma. Patients with a history of CVD without evidence of active disease are eligible for enrollment at the discretion of the study PI.
* Patients with inflammatory bowel disease and/or GI ulcers and/or GI fistulas are eligible but only at the discretion of the study PI after personalized review of their medical history and proximity of SBRT targets to gastrointestinal mucosa.
* Patients with a separate non-cutaneous cancer diagnosis for which the patient has not been without evidence of disease for at least 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | After the completion of SBRT treatment through 3 months of followup.
  This will be accomplished using the standard 3+3 dose escalation design. Dose Limiting Toxicities (DLTs) will be determined through the NCI CTCAE version 4.03.

SECONDARY OUTCOMES:
One Year Local Control | After the completion of SBRT treatment, throughout followup, or death, whichever comes first, up to one year.
  Local Control will be defined as Stable Disease (SD), Partial Response (PR) or Complete Repsonse (CR) according to RECIST 1.1 criteria. Assessed using Kaplan Meier survival curves.
Progression Free Survival | After the completion of SBRT treatment, throughout followup, or death, whichever comes first, up to one year.
  The amount of time a patient survives without worsening of disease, according to RECIST 1.1 criteria. Assessed using Kaplan Meier survival curves.
Overall Survival | After the completion of SBRT treatment, throughout followup, or death, whichever comes first, up to one year.
  The amount of time a patient survives, with or without progression of disease. Assessed using Kaplan Meier survival curves.
Chemotherapy-Free Interval | After the completion of SBRT treatment throughout followup to the re-initiation of chemotherapy, up to one year.
  The amount of time a patient survives without having to undergo re-initiation of chemotherapy. Assessed using Kaplan Meier survival curves.
Acute Toxicities | During SBRT treatment, throughout followup, or death, whichever comes first, up to 6 weeks post treatment.
  Acute toxicities will be assessed by the NCI CTCAE version 4.03.
Late Toxicities | After the completion of SBRT treatment, throughout followup, or death, whichever comes first, up to one year.
  Delayed toxicities will be assessed by the NCI CTCAE version 4.03.
Quality of Life Assessment through Survey | After the completion of SBRT treatment, throughout followup, or death, whichever comes first, up to one year.
  Quality of life will be assessed through the EORTC QLQ-C30 and OV28 questionnaires.
Functional Imaging | Prior to completion of SBRT, immediately after the completion of SBRT, and 6 weeks after the completion of SBRT.
  DCE-CT scans using the Siemens AS open scanner will be assessed according to RECIST 1.1 criteria.
Profile of SBRT-Associated Immune Response | Prior to completion of SBRT, 2 weeks after the completion of SBRT, and 6 weeks after the completion of SBRT.
  The Human Immune Monitoring Shared Resource will preform cytometry and cytokine arrays, as well as characterizing activation markers.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Fisher, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Derived] Robin TP, Hu J, Jones BL, Patton T, Diamond JR, Behbakht K, Lefkowits C, Corr BR, Fisher CM. Phase I trial of stereotactic body radiation therapy (SBRT) for limited site locoregional recurrences of ovarian cancer. Gynecol Oncol. 2025 Sep;200:175-179. doi: 10.1016/j.ygyno.2025.07.023. Epub 2025 Aug 20. PMID 40839922